CLINICAL TRIAL: NCT06710132
Title: PROCEADE PanTumor: A Phase 1b/2, Multicenter, Open-Label Study of Anti-CEACAM5 Antibody-Drug Conjugate M9140 in Participants With Advanced Solid Tumors (Master Protocol)
Brief Title: Study of Anti-CEACAM5 ADC M9140 in Participants With Advanced Solid Tumors (PROCEADE PanTumor)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry); Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS202329_0010; 2024-517817-34-00 (Other: CTIS); 2024-517818-15-00 (Other: CTIS); 2024-517819-74-00 (Other: CTIS)
Record Dates: First submitted 2024-11-22; First posted 2024-11-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors; Gastric Cancer; Non-Small Cell Lung Cancer (NSCLC); Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma (PDAC)
Keywords: ADC; TOP1 inhibitor; Gastric Cancer; Gastroesophageal junction cancer; Non-Small Cell Lung Cancer; Pancreatic Cancer; Solid Tumors
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Substudy GC: M9140 Monotherapy - Part A CEACAM5 High (Experimental)
  Interventions: Drug: M9140
- Substudy GC: M9140 Monotherapy - Part B CEACAM5 Low (Experimental)
  Interventions: Drug: M9140
- Substudy NSCLC: M9140 Monotherapy - Part A CEACAM5 High EGFR Wt (Experimental)
  Interventions: Drug: M9140
- Substudy NSCLC: M9140 Monotherapy - Part B CEACAM5 High EGFR mut (Experimental)
  Interventions: Drug: M9140
- Substudy PDAC: M9140 Monotherapy - Part A CEACAM5 High (Experimental)
  Interventions: Drug: M9140

INTERVENTIONS:
Drug: M9140 — All participants will receive 2.8 milligram per kilogram (mg/kg) M9140 intravenously (i.v.) every 3 weeks (q3w) on Day 1 of consecutive 21-day cycles.
  Other Names: Precemtabart tocentecan

SUMMARY:
The PROCEADE PanTumor study aims to investigate M9140 in multiple tumor types which express carcinoembryonic antigen-related cell adhesion molecule 5 (CEACAM5) and it is therefore designed as a matrix study. This study aims to assess the antitumor activity, tolerability, safety, and pharmacokinetics (PK) of M9140 as monotherapy or in combination treatments in adult participants with locally advanced/metastatic CEACAM5 expressing tumors. There will be 3 substudies under this Master Protocol that may be conducted in parallel.

* PROCEADE PanTumor: A Phase 1b/2, Multicenter, Open-Label Study of Anti-CEACAM5 Antibody-Drug Conjugate M9140 in Participants with Advanced Gastric Cancer (Substudy GC);
* PROCEADE PanTumor: A Phase 1b/2, Multicenter, Open-Label Study of Anti-CEACAM5 Antibody-Drug Conjugate M9140 in Participants with Advanced Non-Small Cell Lung Cancer (Substudy NSCLC);
* PROCEADE PanTumor: A Phase 1b/2, Multicenter, Open Label Study of Anti-CEACAM5 Antibody-Drug Conjugate M9140 in Participants With Advanced Pancreatic Cancer (Substudy PDAC).

DETAILED DESCRIPTION:
The study follows a master protocol concept with several separate substudies in specific indications.

* Substudy GC: The study duration per participant is on an average approximately 10 months. This includes a 28-day Screening period, infusion (approximately 1 hour) on Day 1 of every cycle, and Safety Follow-up Visit 30 (± 3) days after the last dose of M9140.
* Substudy NSCLC: Study duration per participant is approximately 12 months. This includes a 28-day Screening period, infusion (approximately 1 hour) on Day 1 of every cycle, and Safety Follow-up Visit 30 (± 3) days after the last dose of M9140.
* Substudy PDAC: Study duration per participant is on an average approximately 8 months. This includes a 28-day Screening period, infusion (approximately 1 hour) on Day 1 of every cycle, and Safety Follow-up Visit 30 (±3) days after the last dose of M9140.

ELIGIBILITY:
Inclusion Criteria:

* Participants are capable of signing informed consent as defined in protocol
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) below or equal to 1
* Participants with adequate hematologic, hepatic and renal function as defined in protocol
* Participant must have at least 1 lesion that is measurable using RECIST v1.1.
* Other protocol defined inclusion criteria could apply

Substudy GC:

* Participants in Part A and Part B with documented histopathological diagnosis of advanced or metastatic, HER2 negative, gastric or GEJ (with an epicenter 2 centimeter (cm) proximal or distal to the GEJ) adenocarcinoma, who were intolerant/refractory to or progressed after systemic therapies for the advanced/metastatic stage that must have included (provided there is no medical contraindication and these agents are locally approved and available) a fluoropyrimidine and a platinum agent and an Immune checkpoint inhibitors (ICI) for participants with a known microsatellite instability-high (MSI-H) status or participants whose tumor express PD-L1 with a CPS greater than or equal (>=) 1
* Participants must have received and progressed (according to RECIST 1.1) on at least 1 line of therapy for the treatment of advanced/metastatic disease but no more than 2
* Participants in Part A with CEACAM5high GC/GEJC (defined as IHC >= 2+ staining in >= 50% of tumor cells)
* Participants in Part B with CEACAM5low GC/GEJC (defined as IHC >= 2+ staining in less than (<) 50% of tumor cells)
* Other protocol defined inclusion criteria could apply

Substudy NSCLC:

* Participants in Part A and Part B with histologically or cytologically documented advanced (Stage III not eligible for resection or curative radiation) or metastatic NSCLC with or without driver genomic alterations
* Participants must have been intolerant/refractory to or progressed after systemic therapies for the advanced/metastatic stage
* Participants must have received and progressed (according to RECIST 1.1) on at least 1 line of therapy for the treatment of advanced/metastatic disease but no more than 3
* Participants who received a platinum-containing regimen or a targeted therapy as (neo)-adjuvant therapy for early-stage disease, if relapse or metastases occurred during or within 3 months after regimen completion, are considered to have received a line of treatment in the advanced setting
* Participants in Part A with CEACAM5 high-expressing EGFR tumors (including participants with any driver genomic alterations other than EGFR mutations
* Participants in Part B with CEACAM5 high known EGFR mutated tumors as assessed according to local clinical practice
* Other protocol defined inclusion criteria could apply

Substudy PDAC:

* Participants with histologically or cytologically confirmed advanced or metastatic PDAC, who were intolerant/refractory to or progressed after systemic therapies for the advanced metastatic stage that must have included (provided there is no medical contraindications, and these agents are locally approved and available; FOLFIRINOX regimen or NALIRIFNOX regimen or Nab-paclitaxel/gemcitabine regimen
* Participants must have received and progressed (according to RECIST 1.1) on at least one 1 line of therapy for the treatment of advanced/metastatic disease but no more than 2
* All participants will be screened using an IHC test to define CEACAM5 expression. Only participants with CEACAM5high expressing tumors will be eligible
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participant has a history of malignancy within 3 years before the date of enrollment (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, benign prostate neoplasm/hypertropia, or malignancy that in the opinion of the Investigator, with concurrence with the Sponsor's Medical Monitor, is considered cured with minimal risk of recurrence within 3 years)
* Participants with known brain metastases, except those meeting the following criteria: Brain metastases that have been treated locally and are clinically stable for at least 4 weeks prior to the start of treatment; No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
* Participants with diarrhea (liquid stool) or ileus Grade > 1
* Participants with active chronic inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease, intestinal perforation) and/or bowel obstruction
* Cardiac arrhythmia, unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] >= II) or a coronary revascularization procedure within 180 days of study entry. Calculated QTc average (using the Fridericia correction calculation) of > 470 milliseconds (ms)
* Cerebrovascular accident/stroke (< 6 months prior to enrollment)
* Other protocol defined exclusion criteria could apply

Substudy GC - Participants with prior therapy with irinotecan

Substudy NSCLC:

- Participants with prior therapy with irinotecan

Substudy PDAC: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2027-12-23 (Estimated); Study Completion 2027-12-23 (Estimated)

PRIMARY OUTCOMES:
Substudies GC/NSCLC/PDAC: Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigators | Time from first study treatment to (planned) final assessment at approximately 48 months

SECONDARY OUTCOMES:
Substudies GC/NSCLC/PDAC: Number of Participants with Adverse Events (AEs) and Treatment Related AEs | Time from first study treatment to (planned) final assessment at approximately 48 months
Substudies GC/NSCLC/PDAC: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigators | Time from first study treatment to (planned) final assessment at approximately 48 months
Substudies GC/NSCLC/PDAC: Number of Participants with Disease Control | At Week 12
Substudies GC/NSCLC/PDAC: Time to Response according to RECIST v1.1 as Assessed by Investigators | Time from first study treatment to (planned) final assessment at approximately 48 months
Substudies GC/NSCLC/PDAC: Progression-free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigators | Time from first study treatment throughout the study duration until progressive disease or death due to any cause, whichever occur first, approximately 48 months
Substudies GC/ NSCLC/ PDAC: Pharmacokinetic (PK) Plasma Concentrations of M9140 | Cycle (C) 1 Day (D) 1 to C3D15, C4D1 and from C8D1 every 4 cycles on D1 until treatment discontinuation (each cycle is of 21 days), assessed up to approximately 12 months
Substudies GC/NSCLC/PDAC: Number of Participants with Anti-Drug Antibodies (ADA) Against M9140 | Predose (C1D1, C3D1, C8D1) and end of study intervention, assessed up to approximately 12 months
Substudy GC: CEACAM5 expression in tumor | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (61):
- United States (11):
  - University of California - Los Angeles - 300208353, Santa Monica, California
  - Providence Medical Foundation, Santa Rosa, California
  - Georgetown University - Lombardi Comprehensive Cancer Center - 1134847, Washington D.C., District of Columbia
  - D&H Cancer Research Center, Margate, Florida
  - Memorial Cancer Institute at Memorial Healthcare System, Pembroke Pines, Florida
  - Prisma Health Cancer Institute, ITOR, CRU, Greenville, South Carolina
  - Baptist Cancer Center, Memphis, Tennessee
  - Baptist Memorial Health Care -Memphis, Memphis, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Texas M. D. Anderson Cancer Center - Partner, Houston, Texas
  - NEXT Virginia, Fairfax, Virginia
- Australia (4):
  - Flinders Medical Centre, Bedford Park
  - Nepean Cancer Care Centre, Kingswood
  - Mater Misericordiae Ltd - PARENT, South Brisbane
  - Macquarie University Hospital - PARENT, Sydney
- Austria (2):
  - Ordensklinikum Linz Krankenhaus der Elisabethinen Linz - Pneumology, Linz
  - LKH - Universitätsklinikum der PMU Salzburg - Innere Med III/Hämatologie und Onkologie, Salzburg
- France (10):
  - Institut Bergonié - Service d'Oncologie Médicale, Bordeaux
  - Centre Georges François Leclerc - Unité de Phase I, Dijon
  - Centre Oscar Lambret - cancerologie generale, Lille
  - Hopital Albert Calmette - CHU Lille - CHU Lille - Institut Coeur Poumon, Lille
  - Hôpital Européen Georges Pompidou - Hématologie Oncologie, Paris
  - Hôpital Saint-Antoine - Oncologie Médicale, Paris
  - ICO - Site René Gauducheau - Service d'Oncologie medicale, Saint-Herblain
  - Hôpital Foch - Service d'Oncologie Médicale, Suresnes
  - Hopital Rangueil - Service d'Oncologie médicale, Toulouse
  - Institut Gustave Roussy - Pathologie Thoracique, Villejuif
- Italy (3):
  - Arcispedale S. Maria Nuova Azienda Ospedaliera di Reggio Emilia - Servizio di Oncologia, Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Dipartimento di Medicina Interna e Scienze Mediche, Roma
  - Azienda Ospedaliero Universitaria Ospedali Riuniti - UOC Clinica di Oncologia Medica, Torrette Di Ancona
- Japan (8):
  - National Cancer Center Hospital, Chūōku
  - Nara Medical University Hospital - Dept of Oncology, Kashihara-shi
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Saiseikai Kumamoto Hospital - 300175708, Kumamoto
  - Kurume University Hospital, Kurume-shi
  - Niigata Cancer Center Hospital - 300176282, Niigata
  - Kindai University Hospital, Osakasayama-shi
  - NHO Hokkaido Cancer Center - 300175802, Sapporo
- South Korea (9):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System - Division of Infectious Diseases, Seoul
- Spain (14):
  - Hospital Universitario Reina Sofia - Dept of Oncology, Córdoba, CÃ³rdoba
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol - Servicio de Oncologia Medica, Badalona
  - Hospital Universitari Vall d'Hebron - Oncology Dept., Barcelona
  - Hospital Clinic de Barcelona - Servicio de Oncologia, Barcelona
  - Hospital HM Nou Delfos - START Barcelona, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals - Servicio de Oncologia, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañon - Servicio de Oncologia Medica, Madrid
  - Centro Integral Oncologico Clara Campal - Unidad de Fase I-Oncologica, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz - START Madrid FJD - Oncology Phase I, Madrid
  - Hospital Universitario Ramon y Cajal - Servicio de Oncologia, Madrid
  - NEXT Madrid - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Virgen Macarena - Oncology Service, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitari i Politecnic La Fe - Oncology Department, Valencia

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: https://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS202329_0010
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html